CLINICAL TRIAL: NCT05486520
Title: A New Breast Cancer MRI Biomarker Using the Intrinsic T1rho Signal
Brief Title: Low-field MRI for Breast Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Matthew S. Rosen, Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-579
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Benign; Malignant Neoplasm of Breast; Breast Malignant Tumor
Keywords: Breast pathologies benign; Breast pathologies malignant
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BREAST MRI IMAGES FROM HEALTHY VOLUNTEERS (Active Comparator): All participants will be recruited prior to their scheduled diagnostic imaging or diagnostic procedures.
  The expected time to complete the study is a maximum of 1.5 hours with approximately 30-60 minutes of scan time, depending on the specific MRI software being tested.
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- BREAST MRI IMAGES FROM PERSONS WITH KNOWN BREAST PATHOLOGIES BENIGN AND MALIGNANT (Experimental): All participants will be recruited prior to their scheduled diagnostic imaging or diagnostic procedures.
  The expected time to complete the study is a maximum of 1.5 hours with approximately 30-60 minutes of scan time, depending on the specific MRI software being tested.
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — MR images will be acquired using an ultra-low magnetic field 6.5 mT scanner located at the Martinos Center. The study time is estimated to be a maximum of 90 minutes with a maximum of 60 minutes of imaging time

SUMMARY:
This research study wants to learn more about improving the attainable image quality for ultra-low field MRI of the breast using new data acquisition methods(also called MRI pulse sequences) and image reconstruction algorithms.

For this pilot study, are testing a new method to image breast cancers at ultra-low magnetic field. The findings from this breast imaging technique will be compared with results obtained from standard mammograms, ultrasounds, MRIs, clinical examinations, and pathology evaluations, when available. The ultra-low field breast MRI performed for this study will be for research purposes and will not be used to guide clinical care.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first-time investigators are examining the use of ultra-low field MRI to image breast cancer.

The purpose of the study is to develop, test and improve new software techniques for our magnetic resonance imaging (MRI) systems. In developing new, ultra-low field MRI scanners develop sequences and other software algorithms from time to time.

This study will enroll both healthy participants and persons with breast cancer. This investigation will also compare these images to standard mammograms, ultrasounds, MRIs, clinical examinations, and pathology evaluations when available.

It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the adult volunteer subjects by the principal investigator, the coinvestigators, or the study staff prior to the imaging session. The investigator obtaining consent will explain in detail the protocol of the study, its purpose, and potential benefits to the society.
* Subjects will be informed about the minimal risks of ultra-low magnetic fields) and of low-frequency nonionizing RF radiation involved in ultra-low field MR imaging. Subjects will also be informed about small space within the magnet. Unlike high-field scanners, there is essentially no sound produced by the imaging gradients, so hearing protection is not required.
* Subjects will be informed that if they feel uncomfortable with the study, they can choose to terminate the study at any time. They will be informed that their refusal to participate in the study or choosing to terminate it at some point will have no effect on care and treatment received by them at MGH now or in future.
* The subjects will be informed that their personal information will be protected as per the HIPAA guidelines.
* The subjects will have at least 15 minutes to consider participation.
* Subjects will undergo MR contraindication screening to ensure that they meet the basic inclusion/exclusion criteria for the study and give written informed consent immediately prior to the MR imaging study.
* Recruit adult female volunteers of any race or ethnic background, between the ages of 20 to 80, who are either scheduled for breast imaging and/or a percutaneous biopsy.
* All efforts will be taken to find interpreters for volunteers who do not understand English, enabling them to be screened and consented with the short-form consent form so that they may participate in this study.

Exclusion Criteria:

* Exclusion criteria include MR contraindications
* Electronic implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* Ferromagnetic objects such as jewelry or metal clips in clothing
* Pregnant or breast feeding women
* A history of uncontrolled seizures
* Claustrophobia
* Any greater than normal potential for cardiac arrest
* Subjects less than 18 years of age or over 80 years of age.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
T1rho dispersion signal | 1 year
  Student's t-test to compare T1rho dispersion: a) in all participants between fat and fibroglandular tissues (expected difference); b) in patients between fat and cancer tissues (expected difference); and c) in patients between fibroglandular and cancer tissues (expected difference in dispersion curve).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Rosen, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation